CLINICAL TRIAL: NCT05971641
Title: The Effect of Progressive Relaxation Exercises on Postoperative Pain Intensity, Sleep Quality, and Recovery in Patients Undergoing Total Knee Arthroplasty
Brief Title: The Effect of Progressive Relaxation Exercises on Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Rumeysa Birkanım, Nurse, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bartın U
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Total Knee Replacement; Progressive relaxation exercises

STUDY DESIGN:
Intervention Model Description: Two group with a progressive relaxation exercise intervention group
Who Masked: Participant
Masking Description: A total of 96 patients will be recruited based on the sample size calculated using G-power analysis. Through block randomization, 48 patients will be assigned to the intervention group and 48 patients to the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The experimental group is the one in which progressive relaxation exercises will be taught, and we will monitor the results in patients.
  Interventions: Other: progressive relaxation exercise
- control group (No Intervention): The control group is the one in which the service routine is implemented, and progressive relaxation exercises are not taught but monitored.

INTERVENTIONS:
Other: progressive relaxation exercise — Patients who undergo total knee replacement surgery in the experimental group will be taught progressive relaxation exercises. The exercise will last for 30 minutes and will be applied twice a day. Patients will wear a smart wristband. Patient Information Form, Numeric Rating Scale, Richard Campbell Sleep Quality Survey, and Postoperative Recovery Index Scale will be administered. The scales will be filled out for 5 days and will take approximately 10-15 minutes.
  Arms: intervention group

SUMMARY:
The indicators of patient recovery in the postoperative period include sleep, physical functionality, mental health, cognitive functionality, pain, and psychosocial functionality.

This thesis aims to investigate the effects of progressive relaxation exercises on postoperative pain intensity, sleep quality, and recovery in patients undergoing total knee arthroplasty.This study, designed as a randomized controlled experimental study, will be conducted between September 1, 2023, and August 1, 2024, at ÇAYCUMA State Hospital in ZONGULDAK province, Turkey, among patients undergoing total knee arthroplasty. A total of 96 patients will be recruited based on the sample size calculated using G-power analysis. Through block randomization, 48 patients will be assigned to the intervention group and 48 patients to the control group. Data will be collected using the Numeric Rating Scale for pain, the Richard-Campbell Sleep Scale, a sleep tracker smart wristband to measure sleep quality and duration, the Postoperative Recovery Index, and a Patient Information Form.

DETAILED DESCRIPTION:
Introduction: Knee osteoarthritis is observed in approximately 6% of adult individuals. Knee osteoarthritis, which causes pain in individuals, often results in the impairment of their daily lives. Total knee arthroplasty surgery is considered as the final method in the treatment process of knee osteoarthritis. The indicators of patient recovery in the postoperative period include sleep, physical functionality, mental health, cognitive functionality, pain, and psychosocial functionality.

Objective: This thesis aims to investigate the effects of progressive relaxation exercises on postoperative pain intensity, sleep quality, and recovery in patients undergoing total knee arthroplasty.

Method: This study, designed as a randomized controlled experimental study, will be conducted between September 1, 2023, and August 1, 2024, at ÇAYCUMA State Hospital in ZONGULDAK province, Turkey, among patients undergoing total knee arthroplasty. A total of 96 patients will be recruited based on the sample size calculated using G-power analysis. Through block randomization, 48 patients will be assigned to the intervention group and 48 patients to the control group. Data will be collected using the Numeric Rating Scale for pain, the Richard-Campbell Sleep Scale, a sleep tracker smart wristband to measure sleep quality and duration, the Postoperative Recovery Index, and a Patient Information Form. The progressive relaxation exercises Compact disc 8 (CD) prepared by the Turkish Psychologists Association will be used for the patients' progressive relaxation exercise training. The data will be analyzed using the Statistical Package for the Social Sciences (SPSS) program. The data will be presented as numbers and percentages, means and standard deviations, and their distribution will be assessed to determine whether parametric or non-parametric tests should be employed for analysis. The data will be evaluated with a significance level of p<0.05 and a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Without diagnosed mental disorders,
* Without visual, hearing, and speech impairments,
* Proficient in Turkish,
* Diagnosed with gonarthrosis and scheduled for total knee replacement,
* No postoperative complications following total knee replacement surgery,
* Literate with an educational level,
* Pain level of 4 or above on the NRS,
* Receiving analgesic treatment according to the clinical protocol,
* Ownership of a mobile device such as a smart phone or tablet capable of accessing internet-based video content with the latest technology from any brand,
* Patients without diagnosed sleep problems will be included in the thesis study.

Exclusion Criteria:

* Illiterate individuals,
* Under the age of 18,
* Having a condition that hinders communication,
* Referred from another center after surgery,
* Pain level of 4 or below on the NRS,
* Developing complications after total knee replacement surgery,
* Receiving analgesic treatment and methods outside of the clinical protocol,
* Not owning a mobile device such as a smart phone or tablet capable of accessing internet-based video content with the latest technology from any brand,
* Having diagnosed sleep problems,
* Having diagnosed mental disorders, will be excluded from the scope of the thesis study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS): | six day
  The numeric rating scale is used to objectively measure pain and evaluate the effectiveness of pain management. It is utilized to determine patients' pain levels and guide treatment plans. In this scale, participants express their pain level with a specific numerical value. Typically, pain intensity is rated on a scale of 0 to 10, where 0 represents no pain and 10 represents the most severe pain. Participants are asked to indicate their pain intensity using a number based on their own experiences and perceptions. For example, a value between 0 and 2 may indicate mild pain, a value between 3 and 5 may indicate moderate pain, a value between 6 and 8 may indicate severe pain, and a value between 9 and 10 may indicate the most intense pain.

SECONDARY OUTCOMES:
Richard Campbell Sleep Questionnaire (RCSQ): | five day
  The Richard Campbell Sleep Questionnaire (RCSQ), developed by Richards (1987), is a 6-item scale that assesses the depth of nighttime sleep, sleep onset latency, frequency of awakenings, duration of wakefulness upon awakening, sleep quality, and noise levels in the environment. Each item is evaluated on a visual analog scale ranging from 0 to 100. Scores between '0-25' indicate very poor sleep, while scores between '76-100' indicate very good sleep. The scale's total score is based on the evaluation of 5 items, excluding the 6th item that assesses the noise level in the environment. As the score increases on the scale, the quality of patients' sleep also improves.
Postoperative Recovery Index Scale (PRIS): | four day
  The Postoperative Recovery Index Scale (PRIS), developed by Butler et al. in 2012, is a scale that can be used within 30 days after surgery. It is suitable for different surgical procedures. PRIS consists of 5 subscales, which are psychological symptoms, physical activities, general symptoms, bowel symptoms, and desire-satisfaction symptoms. The scores of the items within each subscale are summed, arithmetic means are calculated, and subscale scores are determined. For the total score of PRIS, all 25 items are summed, and the arithmetic mean is taken. Higher scores obtained from the index reflect greater difficulties in postoperative recovery, while lower scores indicate easier postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Rumeysa Birkanım, Msc student, Principal Investigator — Bartın Unıversity

IPD SHARING:
Plan to Share IPD: No